CLINICAL TRIAL: NCT02378025
Title: A Multimodal Evaluation of the Comparative Efficacy of Yoga Versus a Patient Centered Support Group for Treating Chronic Pain in Gulf War Illness
Brief Title: Treating Chronic Pain in Gulf War Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter Bayley, Associate Director of Cognitive Neuroscience, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAY0001AGG; W81XWH-14-1-0615 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain; Gulf War Illness; Chronic Illness
Keywords: Chronic Pain; Veterans; Gulf War Illness
MeSH Terms: conditions — Chronic Pain; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Group (Experimental): Postures, meditation, breathing exercises
  Interventions: Behavioral: Yoga Group
- Pain Management Wellness Group (Active Comparator): Behavioral medicine
  Interventions: Behavioral: Pain Management Wellness Group

INTERVENTIONS:
Behavioral: Yoga Group — A 10-week yoga course designed to treat pain.
  Arms: Yoga Group
Behavioral: Pain Management Wellness Group — A 10-week behavioral therapy course designed to treat pain.
  Arms: Pain Management Wellness Group

SUMMARY:
The purpose of this study is to determine whether yoga is effective for the treatment of chronic pain in Gulf War Illness.

DETAILED DESCRIPTION:
Background:

Many military personnel who participated in the Gulf War in 1990-1991 reported negative health consequences subsequent to their deployment. The most prevalent of these health consequences involves a triad of symptoms that include fatigue, pain and cognitive disturbances, commonly referred to as "Gulf War Illness" (GWI). No clear, unifying patho-physiological disease process or effective treatment has yet been identified for GWI. Results from a diverse spectrum of research studies support the view that veterans with GWI are medically ill, but the physiological abnormalities that contribute to their illness are not currently well understood nor sufficiently treated by conventional medicine. While the cause of GWI remains unknown, a potential link between GWI and autonomic nervous system (ANS) dysregulation has been suggested.

Yoga has been suggested to exert its therapeutic effects through adjusting imbalances in the ANS. In addition, yoga has been shown to be clinically effective in treating many of the physical symptoms typically found in GWI, including chronic pain and fatigue. As chronic pain is perhaps the most prevalent and debilitating symptom of GWI, we propose to target pain. Significantly for this application, no improvements in pain have yet been reported in any clinical trial involving GWI. Furthermore, no published studies have investigated yoga as an intervention in GWI.

Objectives:

The primary objective is to investigate yoga for the treatment of chronic pain in veterans with GWI. A secondary objective is to provide veterans with skills in yoga breathing, postures, and meditation that can be used to promote health and well-being.

Hypothesis 1 (primary):

1. The subjective experience of pain, as measured by the Brief Pain Inventory-Short Form, will be reduced at end of treatment in the group given a 10-week yoga treatment program, compared to a pain support group (control).
2. This effect will be sustained across time and will be found at the end of the 24-week post-treatment follow-up.

Hypothesis 2 (secondary):

Yoga will have a beneficial effect on general well-being; thus, compared to the control group, the yoga treatment group will show benefits across a broad range of measures, including quality of life, fatigue, and medication use.

Specific Aims:

1. To assess the efficacy of yoga in reducing chronic pain and determine if the health-related benefits of yoga persist after termination of the treatment program.
2. To obtain symptom-based outcome measures for veterans with GWI (before and after randomization) to assess pain, fatigue, physical functional status and quality of life.

Study Design:

The intervention to be tested is a 10-week yoga treatment program that has been specially designed for the treatment of chronic pain, as experienced by veterans with GWI. One hundred patients will be randomly assigned to one of two treatment groups: group yoga or a pain management wellness group (control). The control group has been carefully designed to control for many features of a yoga intervention. Patients in both groups will attend weekly classes for 10 weeks, followed by 6 months of follow up. Monitoring will include periodic measures of pain, fatigue, quality of life, and ANS function.

Impact:

Despite increasing demand from veterans for yoga and other forms of complementary and alternative treatments, the provision of yoga in veteran healthcare remains sparse. This is due, in large part, to a lack of randomized clinical trials capable of demonstrating the efficacy and safety of yoga for the treatment of conditions such as GWI. Such a demonstration would strengthen the case to offer yoga as a widely-available treatment for pain in GWI and would help promote yoga as part of integrative healthcare. This treatment trial is designed to begin to determine potential mechanisms of pain maintenance in GWI. If yoga leads to improvement in pain outcome, this would support performing a larger clinical trial of yoga for treating pain and other symptoms of GWI.

ELIGIBILITY:
Inclusion Criteria:

* Served in the military in 1990-1991, regardless of deployment.
* History of chronic pain.
* Able to attend weekly visits at the study center for 10 weeks.
* If on a psychotropic medication, the regimen will be stable for at least 4 weeks, prior to entry in the study.

Exclusion Criteria:

* Participation in another clinical trial.
* Unable to visit the study center.
* Unable to stand or walk.

Ages: 42 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bayley, PhD, Principal Investigator — VA Palo Alto Heath Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Allende S, Mathersul DC, Schulz-Heik JR, Avery TJ, Mahoney L, Bayley PJ. Yoga is effective for treating chronic pain in veterans with Gulf War Illness at long-term follow-up. BMC Complement Med Ther. 2023 Sep 13;23(1):319. doi: 10.1186/s12906-023-04145-y. PMID 37704984
- [Derived] Mathersul DC, Dixit K, Avery TJ, Schulz-Heik RJ, Zeitzer JM, Mahoney LA, Cho RH, Bayley PJ. Heart rate and heart rate variability as outcomes and longitudinal moderators of treatment for pain across follow-up in Veterans with Gulf War illness. Life Sci. 2021 Jul 15;277:119604. doi: 10.1016/j.lfs.2021.119604. Epub 2021 May 11. PMID 33984356
- [Derived] Bayley PJ, Schulz-Heik RJ, Cho R, Mathersul D, Collery L, Shankar K, Ashford JW, Jennings JS, Tang J, Wong MS, Avery TJ, Stanton MV, Meyer H, Friedman M, Kim S, Jo B, Younger J, Mathews B, Majmundar M, Mahoney L. Yoga is effective in treating symptoms of Gulf War illness: A randomized clinical trial. J Psychiatr Res. 2021 Nov;143:563-571. doi: 10.1016/j.jpsychires.2020.11.024. Epub 2020 Nov 11. PMID 33218747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yoga Group | Pain Management Wellness Group
Started | 39 | 36
Completed | 26 | 15
Not Completed | 13 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Group | Pain Management Wellness Group | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (7.2) | 52.0 (6.8) | 53.0 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 31 | 26 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 31 | 29 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 16 | 20 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 39 | 36 | 75

OUTCOME MEASURES:

1. Primary Outcome: Pain (Brief Pain Inventory - Short Form) - Pain Severity
Description: Model - estimated change in the Pain Severity subscale of the Brief Pain Inventory - Short Form from baseline to end of treatment. The subscale's minimum score is 0; maximum is 10; more negative change scores indicate greater improvement from baseline to end of treatment
Time Frame: Week 10 minus Week 0
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga Group | Pain Management Wellness Group
Number analyzed (Participants) | 39 | 36
units on a scale | -.87 (2.49) | -.24 (2.40)
Statistical Analysis 1: Comparison: Yoga Group vs Pain Management Wellness Group; Test type: Superiority; p = .25, Mixed Models Analysis

2. Primary Outcome: Pain (Brief Pain Inventory - Short Form) - Pain Interference
Description: Model - estimated change in the Pain Interference subscale of the Brief Pain Inventory - Short Form from baseline to end of treatment. The subscale's minimum score is 0; maximum is 10; more negative change scores indicate greater improvement from baseline to end of treatment.
Time Frame: Week 10 minus Week 0
Population: Note: One participant was not included in this analysis because he discontinued participation in the study before completing this portion of the baseline assessment.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga Group | Pain Management Wellness Group
Number analyzed (Participants) | 39 | 35
units on a scale | -1.60 (2.32) | -.59 (2.36)
Statistical Analysis 1: Comparison: Yoga Group vs Pain Management Wellness Group; Test type: Superiority; p = .08, Mixed Models Analysis

3. Secondary Outcome: Fatigue (6-Minute Walk Test)
Description: Increase from baseline to end of treatment in distance walked during 6-Minute Walk Test. Greater values indicate more increase and therefore a more positive outcome.
Time Frame: Week 0, Week 10
Population: Three participants did not complete this assessment at baseline, therefore 72 participants are included in this analysis.
Measure: Least Squares Mean (Standard Deviation); unit: meters
Arm/Group | Yoga Group | Pain Management Wellness Group
Number analyzed (Participants) | 38 | 34
meters | 46.4 (119.0) | 14.5 (96.7)
Statistical Analysis 1: Comparison: Yoga Group vs Pain Management Wellness Group; Test type: Superiority; p = .04, Mixed Models Analysis

4. Secondary Outcome: Change in Number of Participants Who Used Analgesic Medication
Description: Change in number of participants who self-reported use of analgesic medication(s) from Week 0 to Week 10.
Time Frame: Week 0, Week 10
Population: Week 0 data reflects all participants who responded to the item; some participants left the item blank. Some participants stated that they could not recall all the medications they were taking. Week 10 reflects all participants who completed the Week 10 assessment and answered the item.
Measure: Number; unit: participants
Arm/Group | Yoga Group | Pain Management Wellness Group
Number analyzed (Participants) | 35 | 31
participants
  Used at Week 0 | 2 | 7
  Used at Week 10: number analyzed (Participants) | 32 | 20
  Used at Week 10 | 4 | 5
Statistical Analysis 1: Comparison: Yoga Group vs Pain Management Wellness Group; Test type: Superiority; p = .25, Regression, Logistic

5. Secondary Outcome: Change in Number of Participants Who Used Nonsteroidal Anti-inflammatory Drugs
Description: Change in number of participants who self-reported use of Nonsteroidal Anti-inflammatory Drug(s) from Week 0 to Week 10.
Time Frame: Week 0, Week 10
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Group | Pain Management Wellness Group
Number analyzed (Participants) | 35 | 31
Participants
  Used at Week 0 | 14 | 15
  Used at Week 10: number analyzed (Participants) | 32 | 20
  Used at Week 10 | 12 | 11
Statistical Analysis 1: Comparison: Yoga Group vs Pain Management Wellness Group; Test type: Superiority; p = .22, Regression, Logistic

6. Secondary Outcome: Change in Number of Participants Who Used Opiate Medication
Description: Change in number of participants who self-reported use of Opiate Medication(s) from Week 0 to Week 10.
Time Frame: Week 0, Week 10
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Group | Pain Management Wellness Group
Number analyzed (Participants) | 35 | 31
Participants
  Participants who used opiates at Week 0 | 4 | 4
  Participants who used opiates at Week 10: number analyzed (Participants) | 32 | 20
  Participants who used opiates at Week 10 | 5 | 5
Statistical Analysis 1: Comparison: Yoga Group vs Pain Management Wellness Group; Test type: Superiority; p = .41, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 34 weeks.
Arm/Group | Yoga Group | Pain Management Wellness Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36
Other Adverse Events (participants affected / at risk) | 0/39 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT02378025/Prot_SAP_000.pdf